CLINICAL TRIAL: NCT03933917
Title: Effect of Large Volume Acute Normovolemic Hemodilution on Perioperative Blood Transfusion and Outcomes in Cardiac Valve Surgery
Brief Title: Application of Large Volume Acute Normovolemic Hemodilution in Cardiac Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-056
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Valve Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Large Volume Acute Normovolemic Hemodilution (Experimental): All the participants will undergo Large Volume Acute Normovolemic Hemodilution.
  Interventions: Procedure: Acute Normovolemic Hemodilution

INTERVENTIONS:
Procedure: Acute Normovolemic Hemodilution — Following induction of anesthesia, the volume of blood to be removed during Acute Normovolemic Hemodilution was calculated using an established formula:V=Weight（Kg）×12-15（mL/Kg）;Blood to be removed was capped at： Vmax=EVB×(Hi-Hf)/Hav（EBV= estimated blood volume （male:70mL/Kg，female:65mL/Kg）；Hi= initial hemoglobin ；Hf=target Hb（ 10g/dL ）；Hav= the average of the initial and minimal allowable hemoglobin）.Ensure the volume of removed blood does not exceed the upper limit and Hb ≥10g/dL after blood removed.

SUMMARY:
The application of acute Normovolemic Hemodilution in cardiac surgery can effectively reduce perioperative blood transfusion, reduce postoperative complications and mortality, and is a low-cost, operable and effective blood protection measure.For the application of Acute Normovolemic Hemodilution in heart surgery, we still face an urgent problem: to what extent can Acute Normovolemic Hemodilution achieve better "blood saving effect", that is, whether a large number of Acute Normovolemic Hemodilution can reduce perioperative blood transfusion to a greater extent.

ELIGIBILITY:
Inclusion Criteria:

1. Audlt patients ( ≥ 18 years old);
2. elective valve surgery under cardiopulmonary bypass;
3. Preoperative hemoglobin (Hb) ≥ 12g/dl; (4) Transfusion Risk Understanding Scoring Tool (TRUST) ≥ 2 (possibility of blood transfusion ≥40%).

Exclusion Criteria:

（1）Low body weight (male: <50 kg;Female: < 45kg);（2）preoperative shock；（3）myocardial infarction within 3 months before surgery；（4）ischemic heart disease;Left main coronary artery stenosis >70%;Severe aortic stenosis (area < 0.7cm2);Severe changes in left ventricular function (ejection fraction <30%, requiring vasoactive agents to assist circulation);（5）uncontrolled hypertension;（6） severe carotid artery stenosis (>70% or with symptoms);（7） kidney failure (blood creatinine level >442 mmol/L) or dialysis treatment;（8） serum albumin level (ALB) is less than 25 g/L.（9） international standardized ratio (INR) >1.5 or platelet count <100 103/mm3;（10）Inherited/acquired coagulation function defect;（11）preoperative preparation platelet;（12） contagious or infectious diseases;（13） patient or family members refused to participate in research;（14）refused to infusion of autologous blood or allogeneic blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Enrollment rate of subjects | Through study completion，about 8 months
  The percentage of patients who completed the study
Completion rate of acute normovolemic hemodilution | Through study completion，about 8 months
  The percentage of patients who complete large volume of acute normovolemic hemodilution
Additional blood transfusion beyond transfusion protocol | Through study completion，about 8 months
  Nonstandard blood transfusion

SECONDARY OUTCOMES:
Rate of perioperative blood transfusion | Through study completion，about 8 months
  The percentage of red blood, fresh frozen plasma and platelet transfusion
Rate of postoperative cardiac complications | Through study completion，about 8 months
  Including myocardial infarction, heart failure, low cardiac output, pericardial tamponade, severe arrhythmia according to physical and laboratory examination
Rate of postoperative pulmonary complications | Through study completion，about 8 months
  Including moderate and massive pleural effusion, respiratory failure, re-intubation according to physical and laboratory examination
Rate of postoperative neurological complication | Through study completion，about 8 months
  Including cerebral hemorrhage, cerebral infarction according to physical and laboratory examination
Rate of postoperative renal complication | Through study completion，about 8 months
  Need renal replacement therapy
Other severe complication | Through study completion，about 8 months
  Including re-operation, re-admission of intensive care unit, multiple organ dysfunction, all cause death according to physical and laboratory examination and medical record

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Study Chair — Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No